CLINICAL TRIAL: NCT02746146
Title: Impact of a Simple Clinical Tool for Increasing Enrollment on a Kidney Transplant Waiting List for Patients Aged Over 70 and Initiating Dialysis
Brief Title: A Simple Clinical Tool for Increasing Enrollment on a Kidney Transplant Waiting List for Patients Aged Over 70 and Initiating Dialysis
Acronym: KITE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PHRC-I/2015/OM-01; 2016-A00464-47 (Other: RCB)
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic dialysis patients (Experimental): The study population consists of patients over 70 (≥) and under 85 years (<) of age with stage 5 chronic renal disease and initiating a first session of chronic dialysis in the Languedoc-Roussillon and Midi-Pyrénées regions. Eligible patients must have a 3 year prognostic mortality score less than (<) 7 points (Dusseux et al. 2015).
  Intervention: Systematic use of a prognostic score
  Interventions: Other: Systematic use of a prognostic score

INTERVENTIONS:
Other: Systematic use of a prognostic score — The prognostic score is given in Dusseux et al 2015. It will be used as soon as possible after the initiation of dialysis.

SUMMARY:
The main objective of this study is to show that the systematic use of a prognostic score as early as possible after the initiation of dialysis in patients over 70 years of age and with a good prognosis at 3 years of dialysis results in an increase in the number of entries on a kidney transplant waiting list at 12 months after the initiation of dialysis.

This prospective assessment is carried out as part of a historico-prospective before-after study in parallel with a survey of changes in national practices over the same time period via a here-elsewhere type study.

Historical data (i.e the. "before" period) will include incident dialysis cases during the calendar years 2013, 2014 and 2015 before the start of the prospective phase (i.e. "after" period, which is represented by the current declaration); since a preliminary study demonstrated that the data are comparable from 2011 to 2013, we will use the average of data thus obtained. Historical data will be retrieved from the REIN (The French Renal Epidemiology and Information Network) registry data and will be validated by investigators at each center.

DETAILED DESCRIPTION:
The secondary objectives are:

A. To show that the systematic use of the score at the initiation of dialysis can shorten the registration delay on a kidney transplant waiting list; to evaluate the time between initiation of dialysis and registration on a national waiting list for kidney transplants, while assessing the duration of the pre-transplant assessment.

B. To identify barriers to registration on the kidney transplant waiting list as well as the related time delay in this population (medical and non-medical factors), the rates and causes of patient refusal for registration and the possible evolution this refusal over time.

C. To evaluate the economic impact of the introduction of the renal transplant clinical prognostic score.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 months of follow-up
* Patient initiating chronic dialysis (incident cases)
* Patients with a 3 year prognostic mortality score less than (<) 10 points (Dusseux et al. 2015)

Exclusion Criteria:

* The patient is participating in another interventional study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Patient on preemptive kidney transplant waiting list (before the initiation of a chronic dialysis program)

Ages: 70 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
The % number of registrants on the kidney transplant waiting list | 12 months

SECONDARY OUTCOMES:
Delay between the initiation of dialysis and inclusion on the kidney transplant waiting list | 12 months
  This outcome integrates the the duration of initial assessment and is measured by the difference between the start and end dates of the pre-transplant assessment.
The number of refusals by patients for registration on the kidney transplant waiting list | 12 months
In case of patient refusal for registration, the reasons why (qualitative approach) | 12 months
The number of cases where there is a medical contra-indication for registration on the kidney transplant waiting list | 12 months
In case of a medical contra-indication for registration on the kidney transplant waiting list, the cause (qualitative approach) | 12 months
The cost of care associated with dialysis patients and dialysed-and-then-transplanted patients will be estimated from the point of view of the French health insurance system | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Moranne, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (25):
- France (25):
  - Clinique Claude Bernard, Albi
  - AIDER - Unité de Dialyse d'Alès, Alès
  - CH d'Auch, Auch
  - Centre d'Hemodialyse Languedoc Méditérranéen, Béziers
  - Medipole Grand Sud St Roch, Cabestany
  - CH de Cahors, Cahors
  - NephroCare, Castelnau-le-Lez
  - CH de Carcassonne, Cité de Carcassonne
  - AAIR Midi-Pyrénées, Colomiers
  - Centre Hospitalier Intercommunal du Val d'Ariège, Foix
  - Clinique du Pont de Chaume, Montauban
  - AIDER de Montpellier, Montpellier
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - Clinique de l'Occitanie, Muret
  - Polyclinique Le Languedoc, Narbonne
  - AIDER - Unité de Dialyse de Nîmes, Nîmes
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Gardialyse, Nîmes
  - CH de Perpignan - Hôpital Saint Jean, Perpignan
  - Centre Hospitalier Jacques Puel, Rodez
  - CH de Bigorre, Tarbes
  - CHRU de Toulouse - Hôpital de Rangueil, Toulouse
  - CHRU de Toulouse - Hôpital Larrey, Toulouse
  - CHRU de Toulouse - Hôptal Casselardit, Toulouse
  - Clinique Néphrologique Saint-Exupéry, Toulouse

REFERENCES:
- [Background] Dusseux E, Albano L, Fafin C, Hourmant M, Guerin O, Couchoud C, Moranne O. A simple clinical tool to inform the decision-making process to refer elderly incident dialysis patients for kidney transplant evaluation. Kidney Int. 2015 Jul;88(1):121-9. doi: 10.1038/ki.2015.25. Epub 2015 Feb 11. PMID 25671769